CLINICAL TRIAL: NCT04579705
Title: The Effect of Different Surgical Hand Scrubbing Methods and the Duration of Scrubbing Time on the Bacterial Flora
Brief Title: Surgical Hand Scrubbing Methods and the Duration of Scrubbing Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Emine Arici Parlak, Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 13131313
Record Dates: First submitted 2020-09-21; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Surgical Scrubbing; Surgical Site Infection
Keywords: scrubbing; scrubbing time; bacterial flora; nursing
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It is the blind that makes microbiological and statistical analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Brushed-1 minute) (Experimental): Surgical hand scrubbing will be performed in 1 minute using a brush.
  Interventions: Other: Using a brush
- Group II (Brushless-1 minute) (No Intervention): Surgical hand scrubbing will be performed in 1 minute without using a brush.
- Group III (Brushed-2 minutes) (Experimental): Surgical hand scrubbing will be performed in 2 minute using a brush.
  Interventions: Other: Using a brush
- Group IV (Brushless-2 minutes) (No Intervention): Surgical hand scrubbing will be performed in 2 minute without using a brush.

INTERVENTIONS:
Other: Using a brush — Surgical hand scrubbing will be performed in 1 minute and 2 minutes using a disposable nail brush.
  Arms: Group I (Brushed-1 minute); Group III (Brushed-2 minutes)

SUMMARY:
Surgical hand scrubbing is the removal of transient flora and reduction of permanent flora as much as possible before any sterile gloves are worn before any surgical intervention. It is a cheap and easy method to prevent infections. Effective use of surgical hand scrubbing has an important role in preventing and reducing the transfer of health-related infections. Although many studies have been performed on surgical hand scrubbing, no standard practice has been found in the method of scrubbing and optimal duration of scrubbing time. The aim of this study is to compare evidence-based surgical hand scrubbing methods in order to prevent surgical site infections.

Methods H0: There is no difference between the effectiveness of different surgical hand scrubbing methods on the bacterial flora in the hand H1: There is a difference between the effectiveness of different surgical hand scrubbing methods on the bacterial flora in the hand.

Time H0: There is no difference between the effectiveness of different the duration of scrubbing time on the bacterial flora in the hand.

H1: There is a difference between the effectiveness of different the duration of scrubbing time on the bacterial flora in the hand.

DETAILED DESCRIPTION:
Original Value: Surgical site infections (SSI) are a serious problem due to increased morbidity and mortality, prolonged hospitalization, hospitalization and consumption of health resources. It is reported from guides that the several factors like hair removal, skin antisepsis, prevention of hypothermia, antimicrobial prophylaxis, providing adequate oxygenation applied in intraoperative period reduce SSI. In addition to these factors, it is known that hand antisepsis of the surgical team is one of the most important factors in preventing SSI. Surgical hand scrubbing is the removal of transient flora and reduction of permanent flora as much as possible before any sterile gloves are worn before any surgical intervention. It is a cheap and easy method to prevent infections. Effective use of surgical hand scrubbing has an important role in preventing and reducing the transfer of health-related infections. Therefore, the research topic is directly related to patient safety and is considered to be one of the important areas of health services at national and international level in terms of establishing institutional culture in the prevention of surgical site infections. Although many studies have been performed on surgical hand scrubbing, no standard practice has been found in the method of scrubbing and optimal duration of scrubbing time. The aim of this study is to compare evidence-based surgical hand scrubbing methods in order to prevent surgical site infections.

Method: The research is a randomized controlled prospective study. The universe of the research was surgeon and operating room nurses in Gulhane Training and Research Hospital. The sample size is at least 180 people for one-way analysis of variance with G * Power version 3.1.19 software to determine a medium level (0.25) effect size between 4 groups at 0.80 power and 0.05 type I error level calculated (Tsai, 2016). Participants was divided into 4 groups by randomization method.

The participants in the first group performed the surgical hand scrubbing for 1 minute and with using a nail brush.

The participants in the second group performed the surgical hand scrubbing for 1 minute and without using a nail brush.

The participants in the third group performed the surgical hand scrubbing for 2 minute and with using a nail brush.

The participants in the fourth group performed the surgical hand scrubbing for 2 minute and without using a nail brush.

Standard Practices in All Groups

* The application will take place during the first surgeries entered in the morning.
* All groups will be used hand antiseptic (4% Chlorhexidine gluconate) which is used in the operating room.
* It will be examined whether the nails are smaller than 2 mm. If the nails are long, individuals will be asked to cut their nails with the help of disposable nail scissors before surgical hand scrubbing.
* There will be no nail polish on the nails and there will be no jewelry on the hand and the ring.
* 3 ml of antiseptic solution will be used at each washing stage.

Volunteers' Exclusion Criteria (Different from Exclusion Criteria):

* Participants want to leave the research
* Expected surgery time is less than 1,5 hours.
* A tear / puncture in the glove during the operation.
* During the operation, data collection will be terminated in cases where the sterility of the glove is impaired.

This research will take place in three stages. At all stages (before surgical hand scrubbing, immediately after and at the end of the surgery), culture will be taken from the active hands of the participants with the Glove Juice Method. At all stages, culture will be taken from the participants via Glove Juice Method.

Glove Juice Method It is a method used to determine the number of bacteria on hand. In this method, individuals will be provided to wear gloves on their dominant hand. Powder-free sterile gloves were used for all sampling. Then, 50 ml of 'Tryptic Soy Broth' medium was placed inside the glove and all surfaces of the gloved hand were massaged for 60 seconds by the researcher. A sample was taken from the liquid in the glove using aseptic techniques and analyzed.

Applications in Medical Microbiology Laboratory Before surgical hand scrubbing, samples taken with glove liquid technique were diluted 1:10 in Müller Hinton Broth broth in the laboratory (500 μl sample, 4.5 ml. Müeller Hinton Broth). And 300 μl of it was placed on 5% sheep blood agar plates with sterile micropipettes. 1 ml each of the other samples (after surgical hand scrubbing and at the end of the surgery) was spread diluted into three 5 % sheep blood agar plates with sterile micropipettes. All samples were incubated at 35° C for 48 hours under atmospheric conditions. Total bacterial load was determined by counting the total colony forming units (CFU) on the plates.

Statistical Method SPSS (Statistical Package for the Social Sciences) Windows Version 22.00 package program will be used in the statistical analysis of the data obtained at the end of the study. Number,%, mean ± standard deviation, median (25% -75%) values will be used in defining the data. Kolmogorov-Smirnov test will be used to evaluate the suitability for normal distribution. In comparative statistics, appropriate tests will be used according to the normal distribution of the sample. In statistical decisions, p ≤ 0.05 level will be accepted as an indicator of significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Being a surgeon or operating room nurse
* Having six months and more surgical experience
* Agree to participate in the research

Exclusion Criteria:

* Not wanting to participate in the research
* Being allergic to the skin due to surgical antiseptic use
* Being latex allergy
* Wounds and abrasions on the hand and nail edges
* To have used a systematic antibiotic at the data collection stage and within two weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The number of bacteria on hand | ''just before surgical hand scrubbing''
  The effect of brush usage and time on bacterial flora in hand during surgical hand. Bacterial analysis was carried out in three consecutive measurement.
The number of bacteria on hand | 'immediately after surgical hand scrubbing''
  The effect of brush usage and time on bacterial flora in hand during surgical hand scrubbing
The number of bacteria on hand | ''after surgery (between 90-120 minutes after surgical hand scrubbing)''
  The effect of brush usage and time on bacterial flora in hand during surgical hand scrubbing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gulhane Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parlak EA, Iyigun E, Albay A, Bedir O. Impact of methods and duration of surgical hand scrub on bacterial count: A randomized controlled trial. Am J Infect Control. 2021 Nov;49(11):1376-1383. doi: 10.1016/j.ajic.2021.05.006. Epub 2021 May 23. PMID 34029650

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT04579705/Prot_SAP_000.pdf